CLINICAL TRIAL: NCT00325715
Title: AGN 201904 Versus Esomeprazole in the Prevention of Aspirin-induced Stomach or Upper Intestinal Damage in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201904-006
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer | interventions — AGN 201904; Esomeprazole

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AGN 201904
- 2 (Active Comparator)
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: AGN 201904
  Arms: 1
Drug: esomeprazole
  Arms: 2

SUMMARY:
AGN 201904, a proton pump inhibitor, versus esomeprazole in the prevention of stomach or upper intestinal damage following administration of high-dose aspirin in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult Volunteers who have provided written informed consent

Exclusion Criteria:

* Volunteers with a history of upper gastrointestinal disease or who have a current diagnosis of upper gastrointestinal disease.
* Female volunteers who pregnant, nursing, or planning a pregnancy
* Volunteers with a history of drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-04; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Stomach or upper intestinal erosions

CONTACTS AND LOCATIONS:
Locations (1):
- Houston, Texas, United States